CLINICAL TRIAL: NCT05417971
Title: A Phase II Trial of Reduced Intensity Fludarabine and Total Body Irradiation-Based Conditioning Prior to Haplo-Identical Transplantation for Patients With Hematologic Malignancies
Brief Title: Reduced Intensity Fludarabine and TBI Prior to Haplo-Identical Transplantation
Status: Recruiting | Type: Observational
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: NSH 1347
Record Dates: First submitted 2022-05-31; First posted 2022-06-14 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Whole-Body Irradiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fludarabine — Reduced-intensity fludarabine with intermediate-dose TBI
  Other Names: Total Body Irradiation

SUMMARY:
This trial will evaluate the safety and efficacy of RIC HIDT transplant protocol following fludarabine and intermediate-dose TBI 800 cGy utilizing PBSC as the stem cell source.

ELIGIBILITY:
Inclusion Criteria:

* Availability of 3/6 - 5/6 matched related donor with a negative HLA-cross match in the host vs. graft direction willing to donate peripheral blood stem cells
* KPS >/= 70%
* Hematologic malignancy requiring allogeneic transplantation, with a predicted high risk of relapse following non-myeloablative, low intensity conditioning.

Exclusion Criteria:

* Poor cardiac function (LVEF <45%)
* Poor pulmonary function (FEV, FVC, DLCO <60%)
* Poor liver function (bilirubin >/= 2.5mg/dL; AST or ALT >3xULN)
* Poor renal function (creatinine clearance <40mL/min)
* HIV-positive; active HepB or HepC
* Uncontrolled infection
* Pregnant female or not able to practice adequate contraception
* Debilitating medical or psychiatric illness which would preclude their giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients with any hematologic malignancy that requires an allogeneic transplant from a halpo-identical matched related donor
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the time to recovery of circulating neutrophils and platelets of all patients to determine incidence of graft rejection | 30 days after transplant

SECONDARY OUTCOMES:
Number of patients who are still alive as assessed by survival status at certain timepoints after transplant | 36 months after transplant
Number of patients with relapsed disease as assessed by labs, bone marrow biopsies and radiological scans at certain timepoints after transplant | 36 months after transplant
Number of patients with evidence of graft versus host disease as assessed by weekly progress notes after transplant | 36 months after transplant
Number of participants who died in the absence of relapse or progression as assessed by survival status at certain timepoints after transplant | 1 year after transplant
Number of participants with responses to treatment as assessed by labs, bone marrow biopsies and radiological scans at certain timepoints after transplant | 36 months after transplant
Number of participants with treatment-related adverse events as assessed by CTCAE v.5.0 | 90 days after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Scott Solomon, MD, Principal Investigator — BMTGA
Locations (1):
- Caitlin Guzowski, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No